CLINICAL TRIAL: NCT07257276
Title: A 3D-CT-Based Dual-parameter Model for Predicting Difficult Laryngoscopy in Infants With Pierre Robin Sequence: Internal and Temporal External Validation
Brief Title: 3D-CT-Based Prediction of Difficult Laryngoscopy in Infants With Pierre Robin Sequence
Acronym: PRS-3DCT
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Hu Danling, Investigator, Nanjing Children's Hospital
Other Study IDs: NanjingCH-PRS-2025; FYX202360 (Other: Jiangsu Maternal and Child Health Association)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pierre Robin Sequence (PRS); Difficult Laryngoscopy; Airway Management
Keywords: 3D-CT; Quantitative Imaging; Difficult Airway; Infants; Prediction Model; Pierre Robin Sequence
MeSH Terms: conditions — Pierre Robin Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Easy Laryngoscopy Group: Infants with Pierre Robin sequence classified as Cormack-Lehane grade I-II during direct laryngoscopy. This group represents patients with easy laryngoscopic exposure.
- Difficult Laryngoscopy Group: Infants with Pierre Robin sequence classified as Cormack-Lehane grade III-IV during direct laryngoscopy. This group represents patients with difficult laryngoscopic exposure.

SUMMARY:
This study aims to develop and validate a quantitative prediction model using three-dimensional computed tomography (3D-CT) imaging for identifying infants with Pierre Robin sequence (PRS) at risk of difficult laryngoscopy. A dual-parameter model incorporating the oropharyngeal sagittal area (S2) and the distance between the tongue base and the posterior pharyngeal wall (D4) will be established. Internal validation will be performed using data from PRS infants treated between 2023 and 2024, and temporal external validation will be conducted using an independent cohort from 2025.

This study seeks to provide an accurate, non-invasive tool for preoperative airway risk assessment in PRS infants, thereby improving anesthetic safety and clinical decision-making.

DETAILED DESCRIPTION:
This retrospective cohort study includes infants diagnosed with Pierre Robin sequence (PRS) who underwent mandibular distraction osteogenesis at the Children's Hospital of Nanjing Medical University between January 2023 and September 2025. Preoperative three-dimensional computed tomography (3D-CT) scans will be used to measure quantitative airway parameters, including the oropharyngeal sagittal area (S2) and the distance from the tongue base to the posterior pharyngeal wall (D4).

According to Cormack-Lehane grades obtained during laryngoscopy, infants will be classified into easy (grades I-II) and difficult (grades III-IV) exposure groups. Logistic regression will be used to identify independent predictors of difficult laryngoscopy, and a dual-parameter model combining S2 and D4 will be developed. The model's discrimination, calibration, and clinical usefulness will be assessed by receiver operating characteristic (ROC) curve analysis, calibration plots, and decision curve analysis (DCA).

Internal validation will be performed using bootstrap resampling (1000 iterations), and temporal external validation will be conducted using an independent cohort from 2025. The goal of this study is to construct a simple, objective, and reproducible model that can improve preoperative airway risk evaluation and support anesthetic management in PRS infants.

ELIGIBILITY:
Inclusion Criteria:Infants diagnosed with Pierre Robin sequence (PRS) based on mandibular hypoplasia, glossoptosis, and upper airway obstruction.

Undergoing mandibular distraction osteogenesis under general anesthesia.

Complete preoperative 3D-CT imaging data available.

Complete intraoperative laryngoscopic grading recorded (Cormack-Lehane classification).

-

Exclusion Criteria:

* Presence of other craniofacial syndromes (e.g., Treacher Collins syndrome, Goldenhar syndrome).

Incomplete or poor-quality 3D-CT images.

Missing laryngoscopic grading or intraoperative data.

History of airway surgery before CT imaging.

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study included infants diagnosed with Pierre Robin sequence who underwent mandibular distraction osteogenesis under general anesthesia at Nanjing Children's Hospital between January 2023 and December 2025. All participants had complete preoperative 3D-CT imaging and intraoperative laryngoscopic grading records.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of the 3D-CT-based dual-parameter model for difficult laryngoscopy | From preoperative imaging (3D-CT) to intraoperative laryngoscopic exposure
  The primary outcome is the discriminative ability of the 3D-CT-based dual-parameter model (including S2 and D4) to predict difficult laryngoscopy in infants with Pierre Robin sequence. Predictive performance will be assessed using area under the receiver operating characteristic curve (AUC), sensitivity, specificity, and calibration analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- anjing Children's Hospital, Affiliated with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a retrospective study involving patient privacy-sensitive information.